CLINICAL TRIAL: NCT00902551
Title: Comparison of DNA Image Cytometry and Conventional Cytology for Cervical Cancer Screening in China
Brief Title: DNA Cytometry for Cervical Cancer Screening in China
Acronym: DNACIC
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiRong Guo, Nanjing Medical University
Other Study IDs: NMU-200703-FC012; NJFY-2007-12901
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Cervical Cancer
Keywords: DNA cytometry; Cytology; Diagnosis accuracy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical samples were taken through cervical brush. Feulgen method is used to determine the amount of DNA.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Subjects underwent cervical sample DNA image cytometry
- 2: Subjects underwent cervical sample conventional cytology

SUMMARY:
Very few screenings of any kind will be possible during a woman's lifetime in most low-resource regions, where 80% of the half-million global cases of cervical cancer occur every year. Although a single round of human papillomavirus (HPV) testing was associated with a significant decline in the rate of advanced cervical cancers and associated deaths, whether other methods like as DNA image cytometry can be used as an more accurate means than others in screening cervical cancer or not is yet to be verified. In addition, the accuracy of both DNA image cytometry and conventional cytology is not well known. The investigators hypothesized that DNA image cytometry was superior in screening cervical cancer than conventional cytology.

ELIGIBILITY:
Inclusion Criteria:

* Currently or had been married
* Not pregnant
* Had an intact uterus with no prolapse
* Had no history of cervical cancer
* Living in China

Exclusion Criteria:

* Not willing to participate or finish the study at any time
* History of cervical surgeries

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy women
Sampling Method: Probability Sample
Enrollment: 25000 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The incidence of cervical cancer. | From the testing performed by the investigator (0h) to one year follow-up period

SECONDARY OUTCOMES:
The rate of death. | One year follow-up period after screening.
The incidence of cervical intraepithelial neoplasia. | From the screening (0h) to one year follow-up period
Cervical inflammation | From the screening (0h) to one year follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Tong H, Shen R, Wang Z, Kan Y, Wang Y, Li F, Wang F, Yang J, Guo X; Mass Cervical Cancer Screening Regimen Group. DNA ploidy cytometry testing for cervical cancer screening in China (DNACIC Trial): a prospective randomized, controlled trial. Clin Cancer Res. 2009 Oct 15;15(20):6438-45. doi: 10.1158/1078-0432.CCR-09-1689. Epub 2009 Oct 13. PMID 19825960